CLINICAL TRIAL: NCT06596499
Title: Clinical Outcomes in Patients with a Novel Fully Magnetically Levitated Left Ventricular Assist Devices：A Multicenter Study
Brief Title: Outcomes of a Novel Magnetically Levitated LVAD: a Multicenter Analysis
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Zhongshan Hospital (Other); Wuhan Asia Heart Hospital (Other); Henan Provincial Chest Hospital (Other); Sichuan Provincial People's Hospital (Unknown); Jiangsu Provincial People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: KS2024086
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Left ventricular assist device; CH-VAD; Outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CH-VAD: All patients implanted with the CH-VAD as the primary device
  Interventions: Device: CH-VAD

INTERVENTIONS:
Device: CH-VAD — The CH-VAD pump is a fully magnetically levitated (maglev), centrifugal continuous-flow blood pump.

SUMMARY:
This multicenter, retrospective cohort study evaluates the clinical outcomes associated with a novel fully magnetically levitated left ventricular assist device (LVAD) in patients with advanced heart failure. Data were collected from seven medical centers in China, involving patients who received the CH-VAD device between June 1, 2022, and June 30, 2024. The study aims to assess short-term and long-term outcomes, including survival, myocardial recovery, and device-related complications.

The CH-VAD is designed with a magnetically levitated rotor to minimize mechanical wear and the risk of thrombosis. Patients included in the study were those with end-stage heart failure, selected based on specific clinical criteria, with the CH-VAD being the primary mechanical circulatory support device. Data were extracted from electronic medical records, including demographic information, clinical characteristics, surgical details, and postoperative outcomes.

Exposure factors analyzed include patient demographics, preoperative conditions, and details of the CH-VAD implantation. The primary endpoints were survival to transplant, myocardial recovery, reoperation to replace the original pump, or heart transplantation within 30 days and at 1 year postoperatively. Secondary outcomes included adverse events such as device thrombosis, stroke, and major bleeding.

Statistical analysis was conducted using Kaplan-Meier survival curves and multivariable regression models to evaluate outcomes. The study was approved by the Institutional Ethics Committee of Anzhen Hospital, with a waiver of informed consent due to its retrospective nature.

This study provides data on the clinical outcomes associated with the CH-VAD, contributing to the understanding of its use in patients with end-stage heart failure.

DETAILED DESCRIPTION:
Introduction Heart failure (HF) is a progressive condition that represents the final stage of various cardiovascular diseases, where the heart can no longer maintain adequate circulation. End-stage heart failure (HF) is associated with refractory symptoms that persist despite optimal medical management, often leading to frequent hospitalizations and a high mortality rate of approximately 50% per year. Globally, the prevalence of HF exceeds 60 million, with 6.4 million individuals suffering from end-stage HF. In China, there are an estimated 13 million HF patients, of which 1 million are in the end-stage category. This stage is marked by the inability of standard medical treatments to stabilize the disease, thus placing a heavy burden on healthcare systems.

The primary therapeutic strategies for end-stage HF are heart transplantation (HTx) and mechanical circulatory support (MCS). HTx remains the gold standard, providing the best outcomes in terms of survival and quality of life; however, it is limited by a severe shortage of donor hearts and the complications related to immunosuppressive therapy. Annually, there are around 6,000 heart transplants performed worldwide, with approximately 700 in China. Mechanical circulatory support, particularly left ventricular assist devices (LVADs), has become a critical alternative to HTx for patients with end-stage HF, offering long-term support (destination therapy, DT), bridge to transplantation (BTT), and bridge to recovery (BTR). LVADs have evolved through three generations, from pulsatile to axial-flow to centrifugal-flow designs, the latter of which includes hydrodynamic, magnetohydrodynamic, and fully magnetically levitated devices. In the United States, LVADs are implanted in approximately 3,000 patients annually, surpassing the number of heart transplants. The FDA has approved their use in patients categorized as INTERMACS levels 1 to 4.

LVAD therapy has evolved substantially over the past decade, particularly with the advent of fully magnetically levitated centrifugal pumps like the HeartMate III. This new generation of devices has been shown in large-scale clinical trials to significantly reduce adverse events such as pump thrombosis, stroke, gastrointestinal bleeding, and mortality when compared to earlier devices, such as the HeartMate II. These advantages make LVADs a life-saving option for a growing number of end-stage HF patients, particularly in settings where HTx is not feasible.

The application of LVADs in China began later than in Western countries but has been expanding rapidly in recent years. To date, four LVADs have received regulatory approval in China, one of which is the CH-VAD (BrioHealth Solutions). The CH-VAD is a compact, fully magnetically levitated centrifugal pump designed for long-term mechanical support in patients with end-stage HF. Its small size and fully magnetically levitated impeller reduce mechanical wear, hemolysis, and thrombus formation, contributing to superior hemocompatibility. The first implantation of the CH-VAD took place in 2017 under compassionate use, marking the start of durable LVAD implantation in China. Since then, over 300 patients have received the CH-VAD, with favorable outcomes reported in early clinical studies.

The CH-VAD features several innovative technical characteristics. It measures 25 mm in thickness and 47 mm in diameter, with a weight of only 186 grams, making it one of the smallest LVADs available, thus facilitating easier implantation and reducing ventricular distortion. Despite its compact size, the CH-VAD contains a 33-mm impeller with long blades, which allows for efficient blood flow at lower rotational speeds. This design minimizes shear stress and turbulence, thereby reducing blood trauma and improving hemocompatibility. The CH-VAD's fully magnetically levitated impeller ensures there is no contact between moving parts, thus eliminating mechanical wear and reducing the risk of thrombosis. The pump's flow characteristics have been optimized to ensure stable hemodynamic support with minimal energy consumption, offering a high degree of pass-through pulsatility and adaptability to changing physiological demands.

The pump also has a unique nose cone structure that smooths the change in flow direction, further minimizing turbulence. The U-shaped secondary flow path is designed to enhance washout and reduce stagnation zones, thus improving the overall biocompatibility of the device. The pump operates at speeds ranging from 1,000 to 4,200 revolutions per minute (rpm), providing a flow rate of up to 10 liters per minute (L/min), ensuring adequate perfusion in a wide range of clinical scenarios. The driveline is thin and flexible, with an outer diameter of only 3.3 mm, which may improve patient comfort and reduce the risk of driveline infections, a common complication in LVAD therapy. The CH-VAD system is powered by either two lithium batteries or a combination of a single battery and AC power, offering operational flexibility. Each battery has a capacity of 5200 mAh, providing 6-8 hours of support on a full charge, with a charging time of approximately five hours.

This multicenter observational study aims to evaluate the clinical efficacy and safety of the CH-VAD in end-stage HF patients when the device is used commercially, providing insights into its safety and effectiveness in real-world applications. This study includes all patients who received CH-VAD implants in a post-market approval setting between June 2022 and June 2024 across seven centers in China.

Methods

1. Device description The CH-VAD pump is a fully magnetically levitated (maglev), centrifugal continuous-flow blood pump. Its motor and maglev components are separated, allowing for optimal use of space within the pump. The pump measures 25 mm thick with a diameter of 47 mm and a weight of 186 grams. the compact size facilitates easier implantation and reduces ventricular distortion. Despite its small dimensions, the device contains a 33 mm impeller with long blades, which allows it to spin at a lower operational speed. This reduces turbulence and blood trauma, and achieves a flatter H-Q curve to enhance hemodynamic responsiveness and pass-through pulsatility.

   The device has unique flow paths designed to improve hemocompatibility. A nose cone structure on top of the central post guides the flow to smoothly change direction. A U-shaped secondary flow path has an optimized gap width to minimize turbulence and enhance washout. The speed range of the pump is from 1000 to 4200 rpm and blood flow up to 10 L/min can be delivered. The superior hemocompatibility and flow characteristics have been demonstrated by computational fluid dynamics, bench tests, and animal studies.

   The device also features a very narrow (3.3-mm outer diameter) and flexible driveline, which may improve patient comfort and potentially decrease the risk of infection. The system is powered by either two lithium batteries or a single battery plus AC power. Each battery, with a capacity of 5200 mAh, can sustain the system for 6-8 hours and reaches a full charge within 5 hours.
2. Study Design The study protocol was approved by the institutional ethics committee approval of Anzhen Hospital with a waiver of informed consent. 75 consecutive patients implanted with the CH-VAD between 1 June 2022 and 30 June 2024 across 7 centers in China were included in this retrospective study. This study was initiated and led by Beijing Anzhen Hospital, affiliated with Capital Medical University, and involved six other medical centers from various provinces in China. These centers include Sichuan Provincial People's Hospital in Chengdu, Henan Chest Hospital in Zhengzhou, Shanghai Chest Hospital in Shanghai, Shanghai Zhongshan Hospital in Shanghai, Asia Heart Hospital in Wuhan, and The First Affiliated Hospital of Nanjing Medical University in Nanjing. The study conforms with the Declaration of Helsinki and the ISHLT Ethics statement.
3. Study Population All patients implanted with the CH-VAD as the primary device in a post-market approval setting were included.
4. Data Collection Clinical data collected from electronic clinical records include demographic information, history of presentation, past medical history,, laboratory results, hemodynamic parameters, echocardiography, surgical details, clinical outcomes, adverse events and readmission information.

   4.1 Clinical characteristics

   The following demographic and clinical characteristics of enrolled participants before the operation will be recorded:
   * Sex
   * Age
   * Height (cm)
   * Weight (kg)
   * Etiology of heart failure (ischemic cardiomyopathy, dilated cardiomyopathy, other causes)
   * Preoperative mechanical circulatory support (ECMO, intra-aortic balloon pump [IABP], Impella)
   * Risk factors for cardiovascular diseases and comorbidities (stroke, arterial hypertension, diabetes mellitus, atrial fibrillation, ventricular arrhythmia)
   * INTERMACS profile
   * NYHA
   * History of cardiac surgery
   * History of cardiac intervention 4.2 Echocardiography Transthoracic echocardiogram (TTE) prior to and after LVAD implantation were performed using commercially available machines. By TTE, the chamber sizes, ventricular function, valve function as well as the device function were reviewed.

   4.3 Hemodynamic Parameters

   The following hemodynamic parameters prior to and after LVAD implantation (from the last measurements before the operation to the enrollment) will be collected from the medical records if available:
   * cardiac output (CO) and cardiac index (CI)
   * central venous pressure (CVP)
   * pulmonary artery pressures (PAP), systolic, diastolic and mean PAP
   * pulmonary capillary wedge pressure (PCWP)
   * pulmonary vascular resistance (PVR) 4.4 Laboratory tests

   Laboratory tests conducted prior to and after LVAD implantation (from the last measurements before the operation to enrollment) will be collected via electronic medical records. The following tests will be reviewed if available:
   * Biochemistry: Sodium, potassium, BUN, creatinine, albumin, bilirubin, liver enzymes
   * Hematology: WBC, Hgb, HCT, PLT
   * Coagulation: PT and INR
   * Cardiac Markers: BNP or NT-proBNP 4.5 Perioperative variables

   The following perioperative variables will be collected from the medical records:
   * Surgical approach
   * Concurrent surgical procedures
   * length of ICU stay
   * length of hospital stay (LOS)
   * total surgery time
   * time on the CPB
   * time on aortic cross-clamp 4.6 Patient Health Status Patients' heart failure symptoms and signs retrieved from electronic medical records before and after (from discharge to enrollment) the surgery.
   * Dyspnea
   * Fatigue
   * Edema grades (1 to 4)
   * Abdominal distension
   * Palpitation
   * Loss of appetite
   * NYHA 4.7 Clinical events and Complications All the clinical events and complications post LVAD implantation to enrollment will be retrieved from medical records and re-adjudicated . Definitions of events as described by the INTERMACS guidelines were employed.
   * Hemolysis
   * Right heart failure
   * Device Failure
   * Major bleeding-VAD implantation related bleeding
   * Major bleeding-Gastrointestinal bleeding
   * Major Bleeding - Other Bleeding
   * Major Infection - MCS related infection
   * Major infection-Non MCS related infection
   * Neurological deficit - ischemic stroke
   * Neurological disorder-Hemorrhagic stroke
   * Neurological disorder-TIA
   * Neurological disorder-Other
   * Renal Insufficiency
   * Arrhythmia-Atrial
   * Arrhythmia-ventricular
   * Respiratory failure
   * Venous Thromboembolism
   * Poor Wound Healing
   * Non-Central Nervous System Arterial Thromboembolism
   * Hepatic insufficiency
   * Hypertension
   * Pericardial effusion
   * Myocardial infarction
   * Aortic valve insufficiency
   * Other 4.8 Readmission Readmission events from the discharge of the index hospitalization to enrollment will be collected. The primary cause and duration of each readmission will be collected and analyzed.
5. Outcomes The short-term primary outcome is a composite of survival to transplant, myocardial recovery, reoperation to replace the original pump or heart transplantation within 30 days or during hospitalization.

   The long-term primary outcome is a composite of survival to transplant, myocardial recovery, reoperation to replace the original pump or heart transplantation at 1 year postoperatively.
6. Statistical Analysis Data will be represented as frequency distributions and percentages. Values of continuous variables will be expressed as mean ± standard deviation and median with interquartile range, as necessary. Continuous variables will be compared using independent samples t-tests or Wilcoxon rank-sum tests, where appropriate. Categorical variables will be compared by means of χ2 tests or Fischer's exact test, where appropriate. To analyze changes in echocardiographic and hemodynamic parameters and laboratory values, McNemar matched-pairs tests will be used to compare preoperative values to postoperative values after matching individual patient data. For all analyses, a p < 0.05 will be considered statistically significant. Kaplan-Meier analysis will be used to calculate survival and other time-to-event outcomes. All data will be analyzed using STATA 29 software (IBM, Armonk, NY) and Prism version 9 (GraphPad Software, San Diego, Calif).

ELIGIBILITY:
Inclusion Criteria:

* All patients implanted with the CH-VAD as the primary device in a post-market approval setting were included.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All decisions to undergo surgery came from the multidisciplinary heart failure team including cardiac surgeons, cardiologists, echocardiography specialists, cardiovascular anaesthesiologists, nurses and other specialists. All patients implanted with the CH-VAD as the primary device in a post-market approval setting were included.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
short-term primary outcome | 30 days
  The short-term primary outcome is a composite of survival to transplant, myocardial recovery, reoperation to replace the original pump or heart transplantation within 30 days or during hospitalization.
long-term primary outcome | 1 year
  The long-term primary outcome is a composite of survival to transplant, myocardial recovery, reoperation to replace the original pump or heart transplantation at 1 year postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No